CLINICAL TRIAL: NCT01293591
Title: Garlic Intake And Biomarkers Of Cancer Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Beltsville Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Janet Novotny, Research Physiologist, USDA Beltsville Human Nutrition Research Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: Garlic Study 2010
Record Dates: First submitted 2011-02-08; First posted 2011-02-10 (Estimated); Last update posted 2017-06-02 (Actual); Status verified 2011-02

CONDITIONS: Healthy Men; Healthy Women
Keywords: Garlic; Cancer biomarkers; Gene expression; Oxidative stress; DNA damage

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Other): 270 kcal White bread with 15 g margarine
  Interventions: Other: Control
- Garlic Treatment (Other): 270 kcal white bread with 15 g margarine and 5 g crushed garlic
  Interventions: Other: Garlic treatment

INTERVENTIONS:
Other: Control — Subjects will consume a garlic-free diet for 10 days. On day 11, subjects will consume 270 kcal white bread with 15 g margarine.
  Arms: Control
Other: Garlic treatment — Subjects will consume a garlic-free diet for 10 days. On day 11, subjects will consume 270 kcal white bread with 15 g margarine and 5 g crushed garlic.
  Arms: Garlic Treatment

SUMMARY:
This study is being done to study the healthful benefits of eating garlic. Previous studies suggest that garlic may help prevent cancer. The investigators are recruiting healthy volunteers to participate in a study to determine the ways in which eating garlic may reduce cancer risk.

DETAILED DESCRIPTION:
A crossover design will be utilized with each participant completing each treatment phase; participants will be randomly assigned to a sequence of dietary treatments. There will be a 17-day washout period in between diet periods. Participants will consume a garlic-free diet for the first 10 days of each diet period. The dietary treatments will be administered on day 11 of each diet period. Dietary treatments will be incorporated into food as follows: 1) 5 g (0.175 oz.) of garlic mixed with 15 g margarine on top of 270 kcal white bread, served as breakfast, or 2) 15 g margarine on top of 270 kcal white bread, served as breakfast.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-80 years

Exclusion Criteria:

* Younger than 40 years old or older than 80 years old
* Use of blood-thinning medications such as Coumadin (warfarin), Dicumarol (dicumarol), or Miradon (anisinidione)
* Presence of kidney disease, liver disease, gout, certain cancers, thyroid disease, gastrointestinal, other metabolic diseases or malabsorption syndromes.
* Have been pregnant during the previous 12 months, are currently pregnant or lactating, or plan to become pregnant during the study
* Follicle stimulating hormone levels above 35 mIU/mL serum
* Type 2 diabetes requiring the use of oral antidiabetic agents or insulin
* History of eating disorders or other dietary patterns which are not consistent with the dietary intervention (e.g., vegetarians, very low fat diets, high protein diets)
* Use of prescription or over-the-counter antiobesity medications or supplements (e.g., phenylpropanalamine, ephedrine, caffeine) during and for at least 6 months prior to the start of the study or a history of a surgical intervention for obesity
* Active cardiovascular disease (such as a heart attack or procedure within the past three months or participation in a cardiac rehabilitation program within the last three months, stroke, or history/treatment for transient ischemic attacks in the past three months, or documented history of pulmonary embolus in the past six months).
* Use of any tobacco products in past 6 months
* Use of oral or IV antibiotics during the month preceding the study or during the study
* Unwillingness to abstain from vitamin, mineral, and herbal supplements for two weeks prior to the study and during the study
* Known (self-reported) allergy or adverse reaction to garlic
* Inability to metabolize garlic
* Unable or unwilling to give informed consent or communicate with study staff
* Self-report of alcohol or substance abuse within the past twelve months and/or current acute treatment or rehabilitation program for these problems (Long-term participation in Alcoholics Anonymous is not an exclusion)
* Other medical, psychiatric, or behavioral factors that in the judgment of the Principal Investigator may interfere with study participation or the ability to follow the intervention protocol

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-07; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Garlic metabolites | Day 11 of each treatment period -- before and 3 hours after treatment
  Garlic metabolites will be measured in blood and urine.
Markers of gene expression | Day 11 of each treatment period -- before and 3 hours after treatment
  Lymphocyte microarray analysis, lymphocyte DNA genotyping. Microarray results will be confirmed by RT-PCR.
DNA damage | Day 11 of each treatment period -- before and 3 hours after treatment
  Comet assay, 8-oxo-dG, histone analysis
Oxidative stress | Day 11 of each treatment period -- before and 3 hours after treatment
  Serum nitrate/nitrite, malondyaldehyde, glutathione, glutathione reductase, glutathione S-transferase, catalase, protein carbonyls, F2-isoprostanes.
Biomarkers of inflammation | Day 11 of each treatment period -- before and 3 hours after treatment
  C-reactive protein (CRP), vascular endothelial growth factor, IL-1, IL-6, TNF-α.

CONTACTS AND LOCATIONS:
Locations (1):
- USDA Beltsville Human Nutrition Research Center, Beltsville, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Charron CS, Dawson HD, Albaugh GP, Solverson PM, Vinyard BT, Solano-Aguilar GI, Molokin A, Novotny JA. A Single Meal Containing Raw, Crushed Garlic Influences Expression of Immunity- and Cancer-Related Genes in Whole Blood of Humans. J Nutr. 2015 Nov;145(11):2448-55. doi: 10.3945/jn.115.215392. Epub 2015 Sep 30. PMID 26423732